CLINICAL TRIAL: NCT01485185
Title: A Randomized, Double Blind, Placebo Controlled Study to Investigate the Effect of Donepezil and Gabapentin Combination on an Experimental Pain Model in Healthy Subjects
Brief Title: Gabapentin and Donepezil Combination on Experimental Human Pain Models
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 115484
Record Dates: First submitted 2011-09-29; First posted 2011-12-05 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Pain, Neuropathic
Keywords: Donepezil; allodynia; Gabapentin; Sural nerve stimulation; Electrical hyperalgesia
MeSH Terms: conditions — Neuralgia; Hyperalgesia | interventions — Gabapentin; Donepezil; gamma-Aminobutyric Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Gabapentin lower dose alone (Experimental): low dose
  Interventions: Drug: Gabapentin lower dose
- Gabapentin higher dose alone (Active Comparator): higher dose
  Interventions: Other: Placebo (Dop)
- Gabapentin in combination with donepezil (Experimental): Gabapentin lower dose and donepezil
  Interventions: Drug: Donepezil; Drug: Gabapentin higher dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo (Gaba)

INTERVENTIONS:
Drug: Gabapentin lower dose — Repeat, oral dose
  Arms: Gabapentin lower dose alone
Drug: Donepezil — Repeat, oral dose
  Arms: Gabapentin in combination with donepezil
Other: Placebo (Dop) — Placebo to donepezil, Repeat, oral dose
  Arms: Gabapentin higher dose alone
Other: Placebo (Gaba) — Placebo to gabapentin, Repeat, oral dose
  Arms: Placebo
Drug: Gabapentin higher dose — Repeat, oral dose
  Arms: Gabapentin in combination with donepezil

SUMMARY:
This study will compare the effects of gabapentin alone, and gabapentin + donepezil given together in two types of experimental electrical pain tests in up to 48 healthy male subjects (after 24 recruited in the first cohort an interim analysis will be performed).

The study is a randomized, double blind, placebo controlled, 3 was cross-over design study with incomplete block design and 4 treatment options. Placebo, gabapentin alone (lower dose and higher dose) or gabapentin (lower dose) with donepezil.

DETAILED DESCRIPTION:
This study will compare the effects of gabapentin alone, and gabapentin + donepezil given together in two types of experimental electrical pain tests which will be conducted on the forearm and the lower leg, in 24 healthy male subjects initially. Gabapentin (a drug for treatment of seizure disorders) is one of the drugs being used for the treatment of pain caused by the damage to the nerves. Donepezil is a treatment to improve memory in patients with Alzheimer's disease. 24 more subjects may be recruited following a formal analysis during the trial (called interim analysis), if required for optimal scientific value. The study consists of 1 screening visit,1 visit to establish the baseline pain recordings before any treatment is given, then 3 treatment sessions, followed by a followup visit. Each treatment session consists of 12 days of dosing at home and 2 inpatient days for dosing and pain tests. Each volunteer takes part in 3 treatment sessions. In total, the study will last 15 weeks for each volunteer. There will be 4 treatment options: placebo, higher dose of gabapentin, low dose of gabapentin, low dose of gabapentin + donepezil. All subjects will receive the last two options and one out of the first two options, in a random order selected by a computer before the study starts; neither the volunteers nor the persons conducting the pain assessments nor the study team will know which treatment the volunteers receive during the visits (known as a randomised, double-blind study). The study will be conducted in a specialist clinical research unit with adequate facilities with regard to safety and compliance. The results of the tests in the study will help to understand the effects of gabapentin and donepezil together to design future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18 and 55 years of age inclusive, at the time of signing the informed consent.
2. Body weight ≥ 50 Kilogram (kg) and BMI within the range 18.5-29.9 Killogram per square meter (kg/m2) (inclusive).
3. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, psychiatric history, psychiatric evaluation, laboratory tests and cardiac monitoring.
4. Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin ≤ 1.5x Upper Limit of Normal (ULN)
5. QT duration corrected for heart rate by Bazett's formula (QTcB) or QT duration corrected for heart rate by Fridericia's formula (QTcF) < 450 milli second (msec).

Exclusion Criteria:

1. The subject has either a previous disease or current medical condition, which as judged by the Investigator, may compromise safety or affect the interpretation of efficacy data.
2. History of known or suspected seizures, including infantile febrile, unexplained significant and recent loss of consciousness or history of significant head trauma with loss of consciousness or a family history (first degree relative) of epilepsy or seizures (fits).
3. Abnormalities in 12-lead Electrocardiogram (ECG)
4. Systolic blood pressure (BP) below 90 or above 160mm Hg, or diastolic blood pressure below 50 or above 100 millimeters of mercury (mmHg).
5. History of sensitivity to any of the study medications
6. History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units. One unit is equivalent to 8 g of alcohol: a half-pint (~240 millil litre [ml]) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
7. A positive pre-study drug/alcohol screen at the screening visit.
8. Excessive caffeine drinkers (~5 or more cups a day) .
9. Excessive smokers (>5 /day)
10. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to screening, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
11. Use of any topical steroid or capsaicin preparations in the previous 30 days to screening, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
12. The subject is needle phobic
13. The subject is unable to tolerate the electrical hyperalgesia model or nerve stimulation, including anxiety or atypical response to the stimulation on the training at the screening visit.
14. The subject does not produce an area of allodynia or hyperalgesia to the electrical hyperalgesia model during the screening session.
15. Subject who, in the investigator/designee's judgement, poses a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behaviour and/or any evidence of suicidal ideation on any questionnaires e.g. type 4 or 5 on the C-SSRS in the last 6 months.
16. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the baseline session in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
17. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 84 day period.
18. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
19. Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-10-11 (Actual); Primary Completion 2012-07-03 (Actual); Study Completion 2012-07-03 (Actual)

PRIMARY OUTCOMES:
Area of pin-prick hyperalgesia | Change from baseline visit to day 14 of treatment sessions
  Change in Area between treatment arms (compared to baseline), measured during the electrical hyperalgesia model using 26 Milli Neuton(mN) von Frey filament
Area of touch-evoked allodynia | Change from baseline visit to day 14 of treatment sessions
  Change in Area between treatment arms (compared to baseline), measured during the electrical hyperalgesia model using a cotton bud

SECONDARY OUTCOMES:
Pain threshold | Change from baseline visit to day 14 of treatment sessions
  Change in threshold between treatment arms (compared to baseline), measured from single electrical stimulation of sural nerve
Ongoing pain intensity rating | Change from baseline visit to day 14 of treatment sessions
  Change in intensity between treatment arms (compared to baseline), measured from 11-point numeric rating scale (NRS) where 0=no pain, 10=maximum pain imaginable
Pain Tolerance | Change from baseline visit to day 14 of treatment sessions
  Change in tolerance between treatment arms(compared to baseline), measured from single electrical stimulation of sural nerve
Pain Temporal Summation | Change from baseline visit to day 14 of treatment sessions
  Change in temporal summation between treatment arms (compared to baseline), measured from repetitive electrical stimulation of sural nerve
Intensity of flare | Change from baseline visit to day 14 of treatment sessions
  Change in intensity between treatment arms (compared to baseline), measured from Laser Doppler imaging evoked by electrical hyperalgesia model

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- [Derived] Boyle Y, Fernando D, Kurz H, Miller SR, Zucchetto M, Storey J. The effect of a combination of gabapentin and donepezil in an experimental pain model in healthy volunteers: Results of a randomized controlled trial. Pain. 2014 Dec;155(12):2510-2516. doi: 10.1016/j.pain.2014.09.003. Epub 2014 Sep 10. PMID 25218827
- See also: Results for study 115484 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115484?search=study&study_ids=115484#rs